CLINICAL TRIAL: NCT03435419
Title: Point of Care Tests for Cutaneous Leishmaniasis: Prospective Evaluation of LoopampTM and CL DetectTM Rapid Test for Cutaneous Leishmaniasis Diagnosis in Afghanistan
Brief Title: Evaluation of Point-of-care Tests for the Diagnosis of Cutaneous Leishmaniasis in Afghanistan
Acronym: CLeishPOCAFG
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: P08020-AFG
Record Dates: First submitted 2018-02-05; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Cutaneous Leishmaniases
Keywords: cutaneous leishmaniasis; RDT; LAMP; PCR
MeSH Terms: conditions — Leishmaniasis, Cutaneous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin samples from cutaneous lesions obtained with a dental broach. Sample stored in lysis buffer accompanying the RDT kit. DNA extracted using commercial kit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: Yes

GROUPS / COHORTS (1):
- CL suspects: Individuals with suggestive signs of cutaneous leishmaniasis presenting themselves at the National Malaria & Leishmaniasis Control Program (NMLCP) Leishmaniasis clinic in Kabul, Afghanistan.
  These will be tested by diagnostic tests under evaluation:
  i) LoopampTM Leishmania Detection Kit is a diagnostic test for Leishmania DNA detection ii) CL DetectTM Rapid Test is a diagnostic test for Leishmania antigen detection And their performance compared against a reference combining microscopy and PCR.
  Interventions: Diagnostic Test: LoopampTM Leishmania Detection Kit; Diagnostic Test: CL DetectTM Rapid Test

INTERVENTIONS:
Diagnostic Test: LoopampTM Leishmania Detection Kit — LoopampTM Leishmania Detection Kit is a diagnostic test for Leishmania DNA detection
Diagnostic Test: CL DetectTM Rapid Test — CL DetectTM Rapid Test is a diagnostic test for Leishmania antigen detection

SUMMARY:
New point-of-care (POC) tests are needed and assessing the performance of these tests for cutaneous leishmaniasis (CL) in Afghanistan may help increasing the number of CL patients with access to accurate diagnosis, and enable prompt treatment. Simpler tests could improve treatment access and benefit patients and communities, by reducing the risk of sequelae and the risk of disease transmission. CLeishPOCAFG aims to advance the diagnosis of CL by using more accurate and field-amenable methods.

DETAILED DESCRIPTION:
The investigators enrolled 274 CL suspects in the study to determine the diagnostic performance of LoopampTM Leishmania Detection Kit and CL DetectTM Rapid Test for CL diagnosis in Afghanistan. The study was conducted at the National Malaria & Leishmaniasis Control Program (NMLCP) Leishmaniasis Clinic in Kabul, Afghanistan.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs compatible with cutaneous leishmaniasis
* Age ≥ than two years old.
* Informed consent obtained and documented.
* Clinical samples can be obtained.

Exclusion Criteria:

* Age less than two years old.
* Failure to obtain and document informed consent.
* Cutaneous leishmaniasis suspects from whom, for any reason, the required clinical samples needed for the study cannot be obtained.
* Patients already receiving CL treatment at the time of enrolment.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CL suspects attending the National Malaria & Leishmaniasis Control Program (NMLCP) Leishmaniasis clinic in Kabul will be invited to enroll the study. Samples from prospective participants will be subjected to standard diagnostic procedure (Giemsa's smear microscopy), as well as PCR (confirmation test to be performed at AMC, The Netherlands) and the two new tests under evaluation, in order to determine the diagnostic accuracy of LAMP and CL Detect.
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2016-04-16 (Actual); Primary Completion 2016-06-22 (Actual); Study Completion 2016-07-18 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of CL Detect RDT and Loopamp Leishmania Detection Kit | Through study completion, an average of 6 months
  Sensitivity and Specificity of the two diagnostic tests

CONTACTS AND LOCATIONS:
Overall Officials: Martijn Vink, MD, MPH, Principal Investigator — HealthNet TPO; Israel Cruz, PhD, Study Director — Foundation for Innovative New Diagnostics

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alvar J, Velez ID, Bern C, Herrero M, Desjeux P, Cano J, Jannin J, den Boer M; WHO Leishmaniasis Control Team. Leishmaniasis worldwide and global estimates of its incidence. PLoS One. 2012;7(5):e35671. doi: 10.1371/journal.pone.0035671. Epub 2012 May 31. PMID 22693548
- [Background] Eroglu F, Uzun S, Koltas IS. Comparison of clinical samples and methods in chronic cutaneous leishmaniasis. Am J Trop Med Hyg. 2014 Nov;91(5):895-900. doi: 10.4269/ajtmh.13-0582. Epub 2014 Sep 15. PMID 25223940
- [Background] Marfurt J, Nasereddin A, Niederwieser I, Jaffe CL, Beck HP, Felger I. Identification and differentiation of Leishmania species in clinical samples by PCR amplification of the miniexon sequence and subsequent restriction fragment length polymorphism analysis. J Clin Microbiol. 2003 Jul;41(7):3147-53. doi: 10.1128/JCM.41.7.3147-3153.2003. PMID 12843055
- [Background] Masmoudi A, Hariz W, Marrekchi S, Amouri M, Turki H. Old World cutaneous leishmaniasis: diagnosis and treatment. J Dermatol Case Rep. 2013 Jun 30;7(2):31-41. doi: 10.3315/jdcr.2013.1135. Print 2013 Jun 30. PMID 23858338
- [Background] Notomi T, Okayama H, Masubuchi H, Yonekawa T, Watanabe K, Amino N, Hase T. Loop-mediated isothermal amplification of DNA. Nucleic Acids Res. 2000 Jun 15;28(12):E63. doi: 10.1093/nar/28.12.e63. PMID 10871386
- [Background] Reithinger R, Dujardin JC, Louzir H, Pirmez C, Alexander B, Brooker S. Cutaneous leishmaniasis. Lancet Infect Dis. 2007 Sep;7(9):581-96. doi: 10.1016/S1473-3099(07)70209-8. PMID 17714672
- [Background] De Silva G, Somaratne V, Senaratne S, Vipuladasa M, Wickremasinghe R, Wickremasinghe R, Ranasinghe S. Efficacy of a new rapid diagnostic test kit to diagnose Sri Lankan cutaneous leishmaniasis caused by Leishmania donovani. PLoS One. 2017 Nov 14;12(11):e0187024. doi: 10.1371/journal.pone.0187024. eCollection 2017. PMID 29135995
- See also: WHO. Control of the Leishmaniases — http://apps.who.int/iris/bitstream/10665/44412/1/WHO_TRS_949_eng.pdf